CLINICAL TRIAL: NCT02327897
Title: Natural History of Asthma With Longitudinal Environmental Sampling
Brief Title: NHALES (Natural History of Asthma With Longitudinal Environmental Sampling)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150058; 15-E-0058
Record Dates: First submitted 2014-12-30; First posted 2014-12-31 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-08

CONDITIONS: Asthma
Keywords: Atopic Asthma; Exposures; Disease Progression; Natural History
MeSH Terms: conditions — Asthma; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asthmatic: study group
- non-asthmatic: controls

SUMMARY:
Background:

- Asthma is a serious clinical and public health problem. Researchers want to collect data to better understand how bacteria and other things in the environment can affect people's asthma.

Eligibility:

- Nonsmoking adults age 18 - 60 who have moderate to severe asthma.

Design:

* Participants will complete a medical history form before the first visit.
* Study visits will include collecting medical history, and conducting physical exam, lung and smoking tests. Participants will give blood, urine, stool, dust, saliva, and sputum samples.
* Participants will take tests that measure their breathing abilities. They will give saliva samples for DNA study. They will get kits to collect stool and dust samples at home. They will fill out surveys.
* Participants will have visits every 6 months for 5 years. They can schedule sick visits, if needed, at no cost to the participant. For all visits, they will have asthma check-ups and get treatment, at no cost to the participant.
* Some participants may take part in a sub-study that includes one 4-hour visit. They will have medical history, physical exam, and lung tests. They will have urine tests to check for pregnancy and tobacco exposure. Then they will have bronchoscopy. For this, an intravenous line will be placed in an arm vein. The nose and throat will be numbed. A flexible fiber-optic tube will be inserted into their airways through the nose. Their airways will be examined and areas of their lung will be washed. A small sample of cells will be taken.

DETAILED DESCRIPTION:
This study will be a prospective, longitudinal, observational, single-center, exploratory, natural history study to collect samples and data that will enable prospective explorations of the interaction between environmental exposures and disease progression over time in moderate-severe atopic asthmatics with persistent disease, and facilitate the formation of mechanistic hypotheses. Environmental and body microbiome samples will be collected and stored from participants for future correlation to effects on asthma symptoms and control.

Samples of blood, urine, DNA, saliva, sputum, stool, and household dust will be collected from approximately 200 participants, as well as quality of life information using asthma symptom questionnaires and, if consented, through the use of home devices. Additionally, samples will be collected from the airways of participants enrolled in the bronchoscopy visit. The samples and survey information collected may be used to explore the microbiological and genetic influences of atopic asthma. Data from the analyses of these samples and survey responses may be evaluated in the context of the environmental exposures, clinical outcomes (symptoms, exacerbations, and quality of life), and response to therapy.

Male and female participants aged 18 to 60 years old with moderate-severe, symptomatic atopic asthma will be enrolled. Participants will be excluded from enrollment if they have a history of chronic obstructive pulmonary disease, cystic fibrosis, non-cystic fibrosis bronchiectasis, pulmonary fibrosis, pulmonary hypertension, emphysema, sarcoidosis, or unstable angina. Additionally, participants will be excluded if they have DVT, pulmonary embolism, class III - IV congestive heart failure, or a malignancy under treatment. Current smokers, and individuals who are allergic to methacholine will not be eligible to enroll. Participants will be enrolled for five years and will receive standard of care asthma therapy as indicated. After the initial screening and baseline visits, participants will return for visits semi-annually and for sick visits as needed. Volunteers participating in the bronchoscopy visit will have an additional single visit after completing the baseline visit.

This cohort of 200 participants will form the basis for future asthma study recruitment, and analysis of collected samples and data. Further expansion of the study beyond five years and 200 participants will be desirable if logistically possible.

ELIGIBILITY:
* Inclusion Criteria

Participants must meet all of the following criteria for enrollment:

* Male or female, 18 to 60 years of age
* Must have clinical evidence of moderate-severe atopic asthma:

  * self-reported symptoms suggestive of asthma (such as wheezing, chest tightness, shortness of breath, cough nocturnal symptoms)

within the past year, and

--*a positive methacholine test confirming diagnosis [provocative concentration causing a 20% fall in forced expiratory volume in 1 second (PC20 FEV1) <16 mg/mL for participants on inhaled corticosteroids and <8 mg/mL for participants not on inhaled corticosteroids] or postbronchodilator FEV1 with at least 12% or 200 mL increase in FEV1 or forced volume vital capacity (FVC) on bronchodilator challenge, and

--no other diagnosis that could explain symptoms.

If there is documentation of a recent methacholine challenge, those results may be used in lieu of conducting a secondary methacholine challenge.

* Permanently resides within 50 miles of the CRU.
* Able to present a valid government issued form of identification for entry to the NIEHS campus
* Able to receive asthma treatment medication(s) via mail
* Willingness to comply with instructions regarding medication regimen, diet, and life style as directed by the investigator that are required per protocol
* Access to a vacuum cleaner with a detachable hose component

  * If a woman is found to be pregnant or breastfeeding at the screening or baseline visit, they may continue their participation in the study but will be excluded from participation in the methacholine challenge and bronchoscopy procedures in this study while pregnant.

Bronchoscopy Visit Inclusion Criterion

In addition to the above inclusion criteria, participants must be able to fast for 6 hours (no food or drink, except a small amount of water if needed to take approved medications) prior to the bronchoscopy visit in order to be eligible for enrollment in the bronchoscopy visit.

Exclusion Criteria

Participants meeting any of the following criteria at screening will not be eligible for enrollment or to continue with study visits:

* Current smoker, significant second-hand smoke exposure (defined by urine cotinine >200 ng/mL at screening), or a history of smoking greater than 5 pack years. Smoking encompasses all inhaled products, including e-cigarettes.
* piCO Smokealyzer value of >11ppm
* History of the following comorbidities: chronic obstructive pulmonary disease, cystic fibrosis (CF), emphysema, non-CF bronchiectasis, pulmonary fibrosis, sarcoidosis, unstable angina, pulmonary hypertension
* Allergy or history of adverse reactions to methacholine
* Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with required study procedures
* Comorbid diseases that affect global health or survival- such as DVT, pulmonary embolism, class III - IV congestive heart failure, or a malignancy under treatment

Bronchoscopy Visit Exclusion Criteria

In addition to the above exclusion criteria, participants meeting any of the following criteria will not be eligible for enrollment into the bronchoscopy visit:

* Pregnancy, as indicated by urine pregnancy test, if of childbearing age and/or ability contraindication
* Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with bronchoscopy
* Bleeding disorders
* Facial deformity, major facial surgery
* Asthma exacerbation or respiratory infection less than or equal to 4 weeks prior to study visit
* Severe persistent asthma, defined as by ATS-ERS criteria.
* Allergy or history of adverse reactions to lidocaine
* Temperature >37.6 (Infinite)C; blood pressure <90/50 mm Hg or >160/100 mm Hg; pulse rate <50 or >100 beats/minute
* Body weight <50 kg (<110 lbs)
* The following abnormal lab values (values obtained during clinical assessment):

  * Platelet count <100,000 per microliters
  * White blood cells count <3000 per microliters
  * Absolute neutrophil count <1000 per microliters
  * Hematocrit <35% for both female and male
  * Prothrombin time (PT) / abnormal international normalized ratio (INR) and partial prothromboplastin time (PTT) based on reference laboratory established reference ranges
  * Serum creatinine >1.4 mg/dL

If a participant is recruited for the Bronchoscopy Visit but does not have current lab values (within 4 weeks), the participant may be asked to return to the CRU for an additional blood draw in order to run the requisite clinical assessments for safety purposes. The participant will be compensated for the additional visit. This is anticipated to be a rare occurrence, as the study team will make all efforts to schedule and complete the bronchoscopy procedure while the lab results are current.

Participants with active bronchospasm on the day of the bronchoscopy will not undergo bronchoscopy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from the population at large, including asthmatic participants who visit the CRU for on-going studies. Participants who have successfully completed other CRU studies may be recruited directly for this study. The study will be registered on clinicaltrials.gov. Local public health departments and other clinics may be contacted for help with recruitment of individuals with moderate to severe atopic asthma. In addition, if needed, the study may be advertised in local media outlets.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
The overall goal is to study the natural history of atopic asthma, focusing on moderate to severe asthma. The primary objective is to collect prospective data and samples for future use to better understand the interaction between environmental ... | End of Study
  Results will be evaluated in the context of the environmental exposures, clinical outcomes (symptoms, exacerbations, and quality of life), and response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It isn t known yet if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-E-0058.html